CLINICAL TRIAL: NCT06992973
Title: Prospective Clinical Study on the Efficacy of the Association of Fractionated SRS and Subsequent Surgery in Patients With Brain Metastases
Brief Title: Efficacy of the Association of Fractionated SRS and Subsequent Surgery in Patients With Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS155/IRE/24
Record Dates: First submitted 2025-03-17; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with brain metastases (Experimental): Patients with single metastatic brain lesions with a diameter ≥ 3 cm symptomatic or asymptomatic or with symptomatic brain lesions ≥ 2 cm < 3 cm that are surgically resectable, without or in the presence of a maximum of 3 small synchronous lesions amenable to radiosurgery treatment, will undergo radiation treatment of 27 Gy in three fractions (9 Gy per fraction) on alternate days; If other lesions are present, up to a maximum of 3 lesions and a total volume of 35 cc, these will be treated with radical stereotactic radiosurgery according to guidelines
  Interventions: Radiation: Treatment based on stereotactic radiosurgery

INTERVENTIONS:
Radiation: Treatment based on stereotactic radiosurgery — Treatment based on stereotactic radiosurgery fractionated within 48-72, followed by surgery for symptomatic brain lesions, amenable to surgical treatment, associated or not with a maximum of 3 additional smaller metastatic brain lesions. The dose will be 27 Gy in three fractions (9 Gy per fraction) on alternate days.
  If other lesions are present, up to a maximum of 3 lesions and a total volume of 35 cc, these will be treated with radical stereotactic radiosurgery according to guidelines.

SUMMARY:
In this study, the possibility of performing a preoperative neoadjuvant radiotherapy dose of 27 Gy fractionated in 3 sessions is explored, to maximize the biological effect of the treatment, in patients affected by solid tumors, in particular lung, breast and melanoma, in which brain metastases have arisen, the incidence of which is constantly increasing in relation to the improvements in oncological therapies and the consequent increase in patient survival. It was demonstrated that postoperative stereotactic radiosurgery with this fractionation was effective in improving local disease control at 1 year compared to single-dose stereotactic radiosurgery (91% vs 77%) and in reducing the risk of radionecrosis for metastatic brain lesions of size.

DETAILED DESCRIPTION:
The treatment of potentially resectable brain metastases in association with preoperative fractionated stereotactic radiotherapy (FSRT) involves the administration of radiation therapy to an intact lesion, with the advantage of presenting fewer uncertainties in terms of target definition and does not require the addition of additional irradiation margins.

Furthermore, the reduction of the dose to healthy brain tissue may lead to a lower risk of inducing subsequent radionecrosis. In fact, the volume of healthy brain tissue irradiated is a recognized predictive factor for the induction of radionecrosis. The overall reduction of treatment times (FSRT + Surgery) with higher compliance by patients and improved logistics. Furthermore, potential advantages consist in the fact that a neoadjuvant radiosurgical treatment can potentially prevent cells scattered during surgery from causing neoplastic leptomeningitis, as these would have already received ablative irradiation. That radiation treatment on a target with an intact vascular supply is potentially more effective because the irradiation bed after surgery is more hypoxic.

It has been observed that over 20% of patients undergoing surgical resection of a metastasis do not undergo the planned radiosurgery due to complications, disease progression or other reasons for delay. The treatment therefore offers the possibility of delivering a higher biological dose with a greater probability of local control and a lower risk of meningeal spread and symptomatic radionecrosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with single metastatic brain lesions with a diameter of ≥ 3 cm symptomatic / asymptomatic or with symptomatic brain lesions ≥ 2 cm < 3 cm that are surgically resectable, without or in the presence of max 3 small synchronous lesions amenable to radiosurgery treatment;
* no urgent surgical indication for neurological symptoms or worsening intracranial hypertension;
* age ≥ 18 years;
* performance status according to the Eastern Cooperative Oncology Group (ECOG) scales ≤ 2;
* Karnfosky Performance Status ≥ 60;
* life expectancy greater than 3 months;
* patients assessed as suitable for surgery (ASA score ≤ 3) and in the absence of contraindications to undergoing brain MRI examination without and with contrast medium;
* ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* contraindications to radiotherapy treatment;
* pregnancy;
* inability to follow the procedures, to fill out the questionnaires;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2029-09-26 (Estimated); Study Completion 2029-09-26 (Estimated)

PRIMARY OUTCOMES:
Local disease control | 24 months
  To evaluate the efficacy of treatment based on Fractionated Stereotactic Radiosurgery followed (within 48-72 h) by Surgery for symptomatic brain lesions (susceptible to surgical treatment) associated or not with a maximum of 3 additional smaller brain metastatic lesions (susceptible to radiosurgical treatment). Local control of the disease after 24 months from treatment by carrying out all the evaluations and analyses that are part of the clinical management of this type of patient and required by the planned radio-surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Telera, Doctor, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy